CLINICAL TRIAL: NCT03834090
Title: Comparison of the Effectiveness of Radial Extracorporeal Shock Wave Therapy and Supervised Exercises in the Treatment of Lateral Epicondylitis: A Randomized Controlled Trial
Brief Title: Effectiveness of Radial Extracorporeal Shock Wave Therapy and Supervised Exercises in Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, MUSTAFA CORUM, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015/369
Record Dates: First submitted 2019-02-05; First posted 2019-02-07 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Lateral Epicondylitis
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rESWT (Experimental): the group receiving rESWT
  Interventions: Device: rESWT
- supervised exercises (Active Comparator): the group receiving supervised exercises
  Interventions: Other: Supervised exercises

INTERVENTIONS:
Device: rESWT — rESWT was administered once per week for 3 weeks using a ShockMaster 500 device with 1.8 bar pneumatic pressure, 10 Hz frequency, with 2000 pulses.
  Arms: rESWT
Other: Supervised exercises — A program including post-isometric relaxation, and progressive resistance exercise (eccentric wrist extension) on the wrist extensors
  Arms: supervised exercises

SUMMARY:
No consensus has yet been built on the treatment of lateral epicondylitis (LE) due to the lack of evidence. Although conflicting results are present, radial extracorporeal shock wave therapy (rESWT) has increasingly been used in the treatment of tendinopathy

DETAILED DESCRIPTION:
ESWT and exercise have beneficial effects on the management of tendinopathies owing to their various mechanisms that showed therapeutic efficacy. Owing to its positive outcomes, extracorporeal shock wave therapy (ESWT) has recently been used in the treatment of musculoskeletal system diseases such as plantar fasciitis, Achilles tendinopathy, calcific rotator cuff tendinopathies, and patellar tendinopathy

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of LE was made in the clinical examination, and the diagnosis was confirmed with the Southampton Diagnostic Criteria of "the presence of epicondyle pain, and epicondyle pain and tenderness on resisted extension of the wrist.
* Patients with symptoms lasting longer than 3 months
* with average pain in the previous week detected as 3 or above on a 10-cm visual analogue scale (VAS)
* who were aged over 18 years

Exclusion Criteria:

* pain in the proximal part of the affected extremity (e.g. shoulder pain, neck pain)
* abnormal neurogenic symptoms (e.g. radicular pain, numbness) on the affected extremity
* presence of posterior interosseous nerve entrapment
* congenital or acquired upper extremity deformities that might affect grip strength
* systemic musculoskeletal system or neurologic disorders
* systemic rheumatologic disease or systemic infection
* presence of malignancy, coagulation disorders, and anticoagulant use
* inserted cardiac pacemaker
* history of surgical treatment on the elbow of the affected extremity
* pregnancy.
* patients who were administered other treatments such as physical therapy or steroid injections in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-02-20 (Actual); Primary Completion 2015-08-15 (Actual); Study Completion 2016-01-15 (Actual)

PRIMARY OUTCOMES:
Change Patient-rated Tennis Elbow Evaluation score | Change from Baseline at 1 month and 3 months after treatment.
  The Patient-rated Tennis Elbow Evaluation is a specific questionnaire designed for the evaluation of the disease-specific pain and function/disability in LE. The scores were calculated separately and as the total PRTEE score, where 0 represented the best score, and 100 represented the worst score. The PRTEE consists of a pain scale with 5 items questioning pain during rest and specific activities (0 represents 'no pain' and 10 represents 'the highest pain'), and a function/disability scale with 10 items evaluating difficulties experienced during specific and daily activities (0 represents 'no difficulty' and 10 represents 'the highest difficulty)

SECONDARY OUTCOMES:
Change Visual Analogue Scale score | Change from Baseline at 1 month and 3 months after treatment.
  The self-evaluation of pain severity during rest and activity in the previous week was calculated using a 10-cm VAS scale
Change Roles and Maudsley Score | Change from Baseline at 1 month and 3 months after treatment.
  The Roles and Maudsley score was used to evaluate pain and activity limitation as classified in four categories: 1 point = excellent, "no pain, complete movement, and complete activity;" 2 points = good, "discomfort from time to time, complete movement, and complete activity;" 3 points = fair, "discomfort after long-duration activity;" and 4 points = poor, "pain that restricts activity".
Change Grip Strength score | Change from Baseline at 1 month and 3 months after treatment.
  Grip strength of the affected upper extremity was calculated using a Hydraulic Hand Dynamometer